CLINICAL TRIAL: NCT06570369
Title: A Phase 1, Single-Center, Double-Blind, Randomized, Placebo-Controlled Study to Explore the Effect of SP-624 on Brain Network Analytics in Cohorts of Healthy Adult Subjects and Subjects With Major Depressive Disorder
Brief Title: A Study to Explore the Effect of SP-624 on Brain Network Analytics in Healthy Adults and Adults With Major Depression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtsei Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-624-103
Record Dates: First submitted 2024-08-17; First posted 2024-08-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Depression; Healthy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-624 (Experimental): SP-624 oral capsule, once daily for 2 weeks
  Interventions: Drug: SP-624
- Placebo (Placebo Comparator): Placebo oral capsule, once daily for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-624 — Oral dose, once daily for 2 weeks
  Arms: SP-624
Drug: Placebo — Oral dose, once daily for 2 weeks
  Arms: Placebo

SUMMARY:
The main goal of this clinical trial is to learn if the active study drug (code name: SP-624) has any effect on the electrical activity of the brain in adult healthy volunteers and in adults with major depression. Another goal of the study is to learn if SP-624 improves memory and learning in adults with major depression. The study will also provide additional information on the safety of SP-624 and how well it is tolerated in adult healthy volunteers and adults with major depression.

Researchers will compare SP-624 to a placebo (a look-alike substance that contains no drug) to see if SP-624 has any effect on study tests.

Study participants will:

Take capsules of study drug (SP-624 or a placebo) once daily for 2 weeks; visit the clinic at Screening, Day 1 (first dose of study drug), and Day 15 (last dose of study drug) for checkups and tests; and have phone call check-ups on Day 7 and about 1 week after the last dose of study drug.

ELIGIBILITY:
Key Inclusion Criteria:

* In generally good health
* Body mass index (BMI) between 18.0 and 40.0 kg/m2
* Willing to comply with the requirements of the study
* For participants with depression: must meet study criteria for moderate to severe major depressive disorder

Key Exclusion Criteria:

* Female who is pregnant or breastfeeding.
* Clinically significant health condition or clinically significant abnormal results on screening health tests
* For participants with depression: presence of exclusionary study criteria for co-morbid psychiatric conditions or medication history.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Brain Network Analytics Profile | At the Day 15 Visit, after approximately 2 weeks of daily dosing with the assigned study intervention
  Brain activity using an electroencephalography (EEG) system during rest and while evoking specific brain activity response will be recorded, and artificial intelligence (AI) based analytics will be performed on the EEG recordings to provide a brain network analytic (BNA) profile for each study participant. The BNA profile at the Day 15 Visit will be compared to the BNA profile at Day 1 pre-dose to evaluate changes in the profile after 2 weeks of daily dosing with the assigned study intervention.

SECONDARY OUTCOMES:
Brain Network Analytics Profile | At the Day 1 Visit, completed on study day 1 after the first dose of the assigned study intervention
  Brain activity using an electroencephalography (EEG) system during rest and while evoking specific brain activity response will be recorded, and artificial intelligence (AI) based analytics will be performed on the EEG recordings to provide a brain network analytic (BNA) profile for each study participant. The BNA profile at Day 1 post-dose will be compared to the BNA profile at Day 1 pre-dose to evaluate changes in the profile after a single dose of the assigned study intervention.
Spatial Working Memory Test | At the Day 15 Visit, after approximately 2 weeks of daily dosing with the assigned study intervention (Participants with Depression Only)
Paired Associates Learning Test | At the Day 15 Visit, after approximately 2 weeks of daily dosing with the assigned study intervention (Participants with Depression Only)
Digit Symbol Substitution Test | At the Day 15 Visit, after approximately 2 weeks of daily dosing with the assigned study intervention (Participants with Depression Only)
Treatment Emergent Adverse Events | Through study completion, an average of 22 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CenExel CNS, Garden Grove, California
  - Alivation Research, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No